CLINICAL TRIAL: NCT03238755
Title: Mechanisms of Cardiac Dysfunction in HIV and the Effect of Statins: a Cardiac MRI Study
Status: Active, not recruiting | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Tomas G. Neilan, MD, Physician, Massachusetts General Hospital
Other Study IDs: 2016P001999
Record Dates: First submitted 2017-08-01; First posted 2017-08-03 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-11

CONDITIONS: HIV Infections
Keywords: HIV; Diastolic Dysfunction; Myocardial fibrosis; Statin
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood, plasma, and serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Statin group: HIV-infected individuals receiving statin therapy for the duration of the study
  Interventions: Other: Cardiac MRI/MRS
- Placebo group: HIV-infected individuals receiving placebo therapy for the duration of the study
  Interventions: Other: Cardiac MRI/MRS

INTERVENTIONS:
Other: Cardiac MRI/MRS — whole blood, plasma, and serum

SUMMARY:
In this study, investigators plan to test whether statins can preserve and/or improve diastolic function among asymptomatic persons with HIV who are on anti-retroviral therapy. Both myocardial fibrosis and myocardial steatosis are thought to contribute to diastolic dysfunction and eventually overt heart failure in HIV. HIV-positive participants will undergo cardiac MRI/MRS imaging studies for the evaluation of myocardial fibrosis and myocardial steatosis prior to initiation of statin or placebo therapy and then two years after initiation of statin or placebo therapy. Traditional markers of cardiovascular (CVD) risk, systemic immune activation/ inflammation, HIV-specific parameters (i.e. CD4 count), and markers of myocardial stretch/injury will be assessed in relation to cardiac MRI/MRS outcomes.

ELIGIBILITY:
Inclusion Criteria:

* New enrollment in the REPRIEVE Trial

Exclusion Criteria:

* clinical diagnosis of HFpEF or HFrEF, by subject report
* standard contraindications to MRI procedure based on MRI Patient Procedure Screening Form - including history of severe allergy to gadolinium

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV-infected subjects on ART from the community
Sampling Method: Probability Sample
Enrollment: 129 (Actual)
Dates: Start 2017-07-31 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2026-04-23 (Estimated)

PRIMARY OUTCOMES:
Extracellular Volume (ECV), a measure of myocardial fibrosis on Cardiac MRI | Two years

SECONDARY OUTCOMES:
Diastolic function on Cardiac MRI | Two years

OTHER OUTCOMES:
Myocardial Inflammation on Cardiac MRI | Two Years
Intramyocardial fat on Cardiac MRI/MRS | Two Years
Diastolic function on Cardiac MRI | Two Years
Visceral Adiposity on MRS | Two Years
Biomarkers (inflammation/ immune markers, hormonal markers) and markers of myocardial stretch | Two Years

CONTACTS AND LOCATIONS:
Locations (4):
- United States (3):
  - VA Medical Center-Los Angeles, Los Angeles, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - UTSW Medical Center, Dallas, Texas
- University of Cape Town, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Neilan TG, Nguyen KL, Zaha VG, Chew KW, Morrison L, Ntusi NAB, Toribio M, Awadalla M, Drobni ZD, Nelson MD, Burdo TH, Van Schalkwyk M, Sax PE, Skiest DJ, Tashima K, Landovitz RJ, Daar E, Wurcel AG, Robbins GK, Bolan RK, Fitch KV, Currier JS, Bloomfield GS, Desvigne-Nickens P, Douglas PS, Hoffmann U, Grinspoon SK, Ribaudo H, Dawson R, Goetz MB, Jain MK, Warner A, Szczepaniak LS, Zanni MV. Myocardial Steatosis Among Antiretroviral Therapy-Treated People With Human Immunodeficiency Virus Participating in the REPRIEVE Trial. J Infect Dis. 2020 Jul 9;222(Suppl 1):S63-S69. doi: 10.1093/infdis/jiaa245. PMID 32645158